CLINICAL TRIAL: NCT05093738
Title: Investigation of the Effect of School Based Cognitive Rehabilitation on Cognitive Skills, Academic Performance and Quality of Life in Refugee Children
Brief Title: The Effect of Cognitive Rehabilitation on Cognitive Skills, Academic Performance And Quality of Life in Refugee Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sümeyye Belhan Çelik, Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20/213
Record Dates: First submitted 2021-09-28; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Cognitive Impairment, Variable
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: This prospective studies that measure the effectiveness of a cognitive rehabilitation intervention. Randomized controlled trials (RCT) are prospective studies that measure the effectiveness of a new intervention or treatment. Participants are recruited and randomly assigned to either the intervention or the comparator group. It is important to ensure that at the time of recruitment there is no knowledge of which group the participant will be allocated to; this is known as concealment. It is examined whether there is any difference in the results of the study intervention and also the intervention and control group are compared.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation Group (Experimental): Refugee Children taking cognitive rehabilitation
  Interventions: Other: Cognitive Rehabilitation
- Control Group (No Intervention): Refugee Children not taking cognitive rehabilitation

INTERVENTIONS:
Other: Cognitive Rehabilitation — In the content of the person-centered intervention program, attention, memory, orientation, praxis (motor planning) training; metacognition (metacognition) training; visual perception; There will be cognitive training for executive functions. The intervention will consist of play activities (games, computer-assisted games) for cognitive skills; The games will be applied in a way that suits the child from simple to complex. Visual perception applications (designing blocks, recognizing and sorting the shapes in the picture, matching opposite shapes etc.); attention practices, memory practices, strategy development, space-time orientation, motor planning, games and metacognitive strategies aimed at developing skills such as planning, organization, working memory, impulse control, time management and awareness, abstract thinking, cognitive flexibility will form our intervention program.
  Arms: Rehabilitation Group

SUMMARY:
Children are the most vulnerable group to be affected by war. The long-term effects of exposure to conflict on children's mental, physical and cognitive development have been documented in the context of war and refugee camps. It has been shown that children who experience war have difficulties in cognitive skills such as attention, learning new information, memory and executive functions. Cognitive skills can ensure a child's school readiness and successful participation in school. Therefore, assessment of children's cognitive performance components can provide a more fundamental understanding of their skills and barriers in school performance. Although there are studies to develop occupational therapy programs in schools for refugee children in the world. No intervention studies specifically aimed at cognitive rehabilitation were found. Therefore, it was aimed to perform cognitive rehabilitation for refugee children and to examine the effects of this on cognitive skills, academic performance and quality of life. The hypotheses on which there is no effect of school-based cognitive rehabilitation approach on cognitive skills, academic performance and quality of life in refugees.

The population of the study will be 34 children (17 studies, 17 controls) between the ages of 12 and 16 who scored 12 points or higher on the Post-Traumatic Stress Scale for Children in Istanbul Secondary School and scored below 21 on the Montreal Cognitive Assessment Scale. Loewenstein Occupational Therapy Cognitive Assessment Scale to assess students' cognitive status; Reading Speed Test and Minnesota Writing Test to assess their academic performance; Pediatric Quality of Life Inventory will be used to assess their quality of life. Refugee children in the study (cognitive rehabilitation intervention) and control groups will be evaluated primarily with the help of these assessment scales, and the individuals in the study group will be given 2 sessions of intervention per week for 10 weeks, with an average of 1 hour per session. At the end of 10 weeks, the participants will be re-evaluated with the help of the same scales and the effectiveness of cognitive rehabilitation will be examined.

DETAILED DESCRIPTION:
The criteria for inclusion of volunteers in the study; Scoring 12 points or more from the Post-Traumatic Stress Reaction Scale for Children, getting a score below 21 from the Montreal Cognitive Assessment Scale, being between the ages of 12-16, having experienced war in their country, being Turkish literate, and volunteering of the child and his/her family to work. The exclusion criteria are; Having a known neurological, developmental or learning disability. The data will be collected by asking our questionnaire and scale questions and by evaluating the cognitive skill components such as the attention test practically. Data collection methods are survey and observation. Quantitative research methods will be used to obtain the data.

Post-traumatic stress level and poor cognitive skills are the parameters that will determine the individuals to be included in the study, and the questionnaires the investigators will use for these are the Post-Traumatic Stress Response Scale for Children and the Montreal Cognitive Assessment Scale. CTSS is used to evaluate specific stress symptoms in individuals who are exposed to violence or trauma. Each child should be evaluated by interviewing the participant about the participant's own reactions to the crisis. This questionnaire has 20 items and scores 7-10, mild post-traumatic stress; 10-12 points, moderate post-traumatic stress; A score of 12 and above indicates severe post-traumatic stress.

Montreal Cognitive Assessment Scale is a scale developed to evaluate mild cognitive impairments and evaluates different cognitive abilities consisting of executive functions, visuospatial skills, memory, language, attention and concentration, abstract thinking, calculation and orientation. The application takes about 10 minutes and the highest total score that can be obtained from the test is 30. Accordingly, scores of 21 and above are considered normal. Refugee children who score below 21 will be included in our study. To evaluate memory function according to this scale; recall from short-term memory, five word learning trials, and delayed recall after five minutes (5 points); to assess visual-spatial skills; Clock Drawing Test (3 points) and 3D cube copying (1 point); to evaluate executive functions; Combining consecutive numbers and letters (such as 1-A, 2-B, 3-C) adapted from the Trail Making Test-B form (1 point), verbal fluency (1 point); to evaluate abstract thinking skills; making similarity between two-item words (2 points); to assess attention, concentration and working memory; sequential subtraction (3 points), determination of the target letter among the read letters (1 point) and counting backwards and forwards (1 each), for language evaluation; Naming three relatively less well-known pictures of animals (lion, rhinoceros, camel) (3 points), repeating two complex sentences paying attention to the syntax (2 points), and time and place orientation questions (6 points) are used to evaluate orientation.

After the individuals included in the investigators' study were selected based on the scales described above, the Loewenstein Occupational Therapy Cognitive Assessment Scale was used to evaluate the cognitive status of the refugee children included; Reading Speed Test and Minnesota Handwriting Test to assess their academic performance; Pediatric Quality of Life Scale will be used to assess their quality of life. After the initial evaluation of the intervention group, it will be taken into cognitive training for 10 weeks and final evaluations will be made at the end of 10 weeks. The control group, on the other hand, will not be given cognitive training for 10 weeks after the first evaluation, and after the final evaluation, the participants' will be given cognitive training for 10 weeks in terms of ethics, after comparison with the intervention group.

the Loewenstein Occupational Therapy Cognitive Assessment Scale was developed to assess basic cognitive abilities in people who have suffered brain damage due to traumatic head injuries, strokes and brain tumors. This scale, which is used to evaluate the cognitive status of people whose cognitive skills are affected for any reason; Orientation, visual perception, spatial perception, motor planning, visual motor organization and thinking ability consisted of six main sections and 26 subtests. The application takes 30-45 minutes. Six main sections of the Loewenstein Occupational Therapy Cognitive Assessment Scale and subtests of these sections will be applied to refugee children whose cognitive skills have decreased due to the effect of exposure to war experience, which the investigators will include in our study. In order to evaluate orientation with this scale, the answers of the individual will be evaluated with a score between 1-4 using four questions for place and time orientation. Four subtests will be used to assess visual perception: visual identification of objects, visual identification of shapes, nested shapes, and object constancy. The answers of the patients will be scored between 1-4 points. For motor planning evaluation, 3 tests will be applied and the patient's performance will be scored with points given between 1-4. Motor imitation, by asking the patient to imitate the 4 movements shown; The use of objects will be evaluated by asking the patient to demonstrate how the various given objects have been used. Copying geometric figures to assess visual motor organization; creating a two-dimensional model by combining the shaped parts in the test booklet; copying the figure in the test booklet with nails on the perforated test board; forming the butterfly shape shown in the test booklet on the test booklet with the 9 pieces given; Scoring will be done by observing the activities of transforming this circle into a clock showing 10:15 by placing the numbers of the clock in a circle given as a hollow. Finally, in order to test the categorization, ordering and logic in order to evaluate the thinking ability, the individual will be asked to group 18 plastic pieces of 3 different shapes and 3 different colors, to sort the 5 picture cards given in a mixed order describing an event, and to describe the event.

Pediatric Quality of Life Inventory consists of physical health, emotional functionality, social functionality and school functionality. One of the general quality of life scales, Pediatric Quality of Life Inventory is a 23-item quality of life scale that is suitable for use in large populations such as schools and hospitals, both healthy and diseased children and adolescents. Items are scored between 0-100. The answer to the question is scored 100 if it is marked as never, 75 if it is marked as rarely, 50 if it is marked as sometimes, 25 if it is marked as often, and 0 if it is marked as almost always. The higher the total Pediatric Quality of Life Inventory score, the better the health-related quality of life is perceived. The most important features of the Pediatric Quality of Life Inventory are that it is short, can be filled in about 5-10 minutes, and is easy to administer and score by the researcher.

For the Reading speed test, which the investigators will use to evaluate the participants' academic performance, the number of words in the text will be divided by the reading time per minute. In addition, children's writing functionality for academic performance will be evaluated with the Minnesota Handwriting Test is one of the standardized, validated and reliable tests that evaluates various parameters of writing. Test, writing; It evaluates six categories of legibility, shape, alignment, size, spacing, and typing speed. In the test application, children; copies this string of words written on the paper onto the marked line just below. In the scoring stage, on the basis of 1/16 inch (0.15 cm) length, all deviations, the proportions between letters and the letters within themselves are evaluated by measuring with a ruler over this length. The lowest score in each category of this test is 0, and the highest score is 34.

After the refugee children in the study (cognitive rehabilitation intervention) and control (non-intervention) groups are evaluated with these assessment scales, cognitive rehabilitation (education) will be applied to the participants in the study group, 2 sessions a week (1 hour per session) for 10 weeks. At the end of 10 weeks, the participants will be re-evaluated and the effectiveness of the treatment will be compared both within the study group and between the study and control groups in terms of children's cognitive skills, academic performance and quality of life parameters.

In the content of the person-centered intervention program, attention, memory, orientation, praxis (motor planning) training; metacognition (metacognition) training; visual perception; There will be cognitive training for executive functions. The intervention will consist of play activities (games, computer-assisted games) for cognitive skills; The games will be applied in a way that suits the child from simple to complex.

CONTRIBUTIONS AND BENEFITS TO BE PROVIDED TO THE CURRENT SCIENTIFIC KNOWLEDGE AND PRODUCTION WITH THE REALIZATION OF THE STUDY The most vulnerable group affected by trauma and war experience is refugee children, and school-based interventions for these children are very limited in our country. This thesis will be a school-based first intervention on cognitive skills that include executive functions such as attention, memory, learning new information and abstract reasoning, which are affected by the exposure of refugee children to conflict.

No studies have been conducted in the world or in our country to examine the effectiveness of a cognitive rehabilitation program that is predicted to facilitate the social adaptation of refugees in our country in the short, medium and long term, by contributing to improving the cognitive functionality, academic performance and quality of life of children. This thesis, which will be carried out, is important in terms of filling this gap in the literature. The findings of this study are aimed to guide health planners and policy makers about school-based intervention approaches to be applied to refugee children who have experienced war and are trying to adapt to a different country.

ELIGIBILITY:
Inclusion Criteria:

* Post-Traumatic Stress Reaction Index for Children score should be taken 12 points
* Montreal Cognitive Assessment Scale score should be taken below 21 points
* being between the ages of 12-16
* having experienced war in their country
* Participants must know Turkish well
* Both the child and the parent must volunteer to participate in the study.

Exclusion Criteria:

* Having a known neurological, developmental or learning disability.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2021-10-25 (Estimated); Primary Completion 2022-01-07 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
Loewenstein Occupational Therapy Cognitive Assessment Scale | 10 weeks
  Loewenstein Occupational Therapy Cognitive Assessment battery is a cognitive screening test which is widely used in occupational health. The application takes 30-45 minutes. Loewenstein Occupational Therapy Cognitive Assessment Scale consists of a total of 26 subtests within 6 areas: Orientation (2 items); Visual Perception (4 items); Spatial Perception (3 items); Motor Praxis (3 items); Visuomotor Organization (7 items); and Thinking Operations (7 items). LOTCA score ranges from 26 to 115 points. Minimum score is 26. Maximum score is 115.

SECONDARY OUTCOMES:
Evaluation of reading speed Minnesota Handwriting Test | 10 weeks
  Reading speed: the number of words in the text/reading time x 60 The higher the number of words per minute, the higher the reading speed.
  Minnesota Handwriting Test: It evaluates the broad category of legibility, shape, alignment, size, spacing, and writing. The lowest score in each category of this test is 0, and the highest score is 34. The higher the total Minnesota score, the better the academic performance is perceived.
Quality of Life Scale for Children | 10 weeks
  Scoring of the 23-item scale is done in 3 areas. First, the total score of the scale, secondly the total score of physical health, and thirdly, the total score of psychosocial health, which consists of calculating the item scores evaluating emotional, social and school functionality, is calculated. Items are scored between 0-100. The answer to the question is 0=100 if it is marked as never, 1=75 if it is marked as rarely, 2=50 if it is marked as sometimes, 3=25 if it is marked as often, 4=0 if it is marked as almost always. The total score is obtained by summing the scores and dividing by the number of items filled in.Minimum score is 100 and maximum score is 0.